CLINICAL TRIAL: NCT04740138
Title: Development of DBT/Parent Training Group Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 11192019.028
Record Dates: First submitted 2021-01-07; First posted 2021-02-05 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Parenting; Emotional Distress

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DBT Skills + Parent Training (Experimental)
  Interventions: Behavioral: Dialectical Behavioral Therapy Skills + Parent Training

INTERVENTIONS:
Behavioral: Dialectical Behavioral Therapy Skills + Parent Training — The DBT/Parent training group intervention is a novel integration of three evidence-based treatments (i.e. DBT Skills, Parent Management Training (PMT), and Emotion Coaching (EC)). The DBT Skills portion of each session follows the DBT Skills Training Manual Second Edition and DBT Skills Training Handouts and Worksheets Second Edition. DBT Skills portions cover the four modules of traditional DBT Skills: mindfulness, distress tolerance, emotion regulation and interpersonal effectiveness.
  PMT portions of the intervention cover: praise, positive interactions and parental attention, reward systems, effective commands, use of consequences, and problem solving. EC portions of the intervention cover: psychoeducation on children's emotional development, teaching children to identify and label emotions, validation of children's emotions, handling children's negative emotions, fostering children's positive emotions and parental modeling of emotion regulation and expression.

SUMMARY:
This treatment development study is aimed at developing and pilot testing a 24-week remotely delivered group intervention that integrates three evidence-based treatments: 1) Dialectical Behavior Therapy (DBT) Skills - targeting adult emotion dysregulation, 2) Parent Management Training (PMT) - targeting parenting behaviors linked to child behavioral dysregulation, and 3) Emotion Coaching (EC) - targeting parental emotion socialization practices linked to child emotion dysregulation.

The aims of the study are to:

1. Evaluate the feasibility of the intervention, specifically with respect to its acceptability and its implementation with 4 families in which a parent has elevated levels of emotion dysregulation and their child has elevated levels of emotion or behavioral dysregulation.
2. Examine change patterns in parent and child mental health and parenting quality using a Single Case Experimental Design (SCED) to evaluate both pre-post and weekly changes in these outcomes.

ELIGIBILITY:
Inclusion Criteria:

* parent must be 18+ years of age
* parent must have at least partial custody of a 3-6 year old child
* neither parent nor child may have any known developmental disability
* parent must be proficient in English
* parent must endorse elevated emotion dysregulation and report their child meets a cutoff for emotional and/or behavioral difficulties.
* parent must have access to the internet and Zoom software

Exclusion Criteria:

* parent with developmental disability
* psychotic disorder
* actively suicidal with an active plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-02-24 (Actual); Study Completion 2021-02-24 (Actual)

PRIMARY OUTCOMES:
Change in parental emotion dysregulation | Baseline up to 24 weeks
  Difficulties with Emotion Regulation Scale (DERS). A 36-item self report measure used to assess adult emotion dysregulation. Items are rated on a scale of 1 to 5, with higher scores indicating higher levels of dysregulation. The measure is comprised of six subscales: lack of emotional awareness, lack of emotional clarity, limited emotion regulation strategies, difficulties with impulse control, difficulties engaging in goal-directed behavior, and nonacceptance of emotional responses.
Change in child behavior | Baseline up to 24 weeks
  Strengths and Difficulties Questionnaire (SDQ). A 25-item parent-report measure in which parents rate (on a Likert scale of 0-2) how characteristic of their child are emotional and behavioral strengths and difficulties. The measure yields a total difficulties score as well as subscales for emotional symptoms, conduct problems, hyperactivity, peer problems and prosocial behavior. Internalizing and Externalizing sub scales can also be generated. Higher scores indicate greater difficulties.
Change in parenting Quality | Baseline up to 24 weeks
  Parenting Scale (PS). A 30-item self-report questionnaire, in which parents are asked to describe (on a Likert scale of 1-7) how they respond to a variety of child misbehaviors. The measure yields three subscales: laxness, over-reactivity and hostile parenting. Higher scores indicate more dysfunctional parenting behaviors.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Oregon, Eugene, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2020-07-27): https://cdn.clinicaltrials.gov/large-docs/38/NCT04740138/ICF_000.pdf